CLINICAL TRIAL: NCT01447654
Title: INHibition of the Renin Angiotensin System in Hypertrophic Cardiomyopathy and the Effect on Ventricular Hypertrophy - a Randomized Intervention Trial With Losartan.
Brief Title: Inhibition of the Renin Angiotensin System With Losartan in Patients With Hypertrophic Cardiomyopathy
Acronym: INHERIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henning Bundgaard (Other)
Responsible Party: Sponsor-Investigator, Henning Bundgaard, Consultant, dr. med., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-001191-19
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic cardiomyopathy; Hypertrophic obstructive cardiomyopathy; Hypertrophy; Losartan; Angiotensin II receptor antagonist
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypertrophy | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Losartan (Active Comparator)
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — 100 mg for 12 months.
  Arms: Losartan
Drug: Placebo — 100 mg for 12 months.
  Arms: Placebo

SUMMARY:
Objective The objective of the study is to assess the structural and functional cardiac effects of treatment with losartan in patients with hypertrophic cardiomyopathy (HCM).

Design The study is a randomized, placebo-controlled, double-blinded trial. The follow-up period is 12 months. 130 patients with HCM will be included in predefined subgroups. Genotype positive relatives with borderline hypertrophy (> 13 mm) will also be included. Data on individuals with borderline hypertrophy will be analysed separately from the rest of the cohort.

Primary outcome Ventricular hypertrophy assessed as left ventricular mass and maximal wall thickness.

ELIGIBILITY:
Inclusion Criteria:

* Hypertrophic cardiomyopathy
* > 18 years
* Sinus rhythm

Exclusion Criteria:

* EF < 50 %
* Treatment with RAS-inhibitor
* Contraindications to losartan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hypertrophy of left ventricle | 12 months
  Left ventricular mass. Maximal wall thickness.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of cardiology, Rigshospitalet., Copenhagen, Denmark

REFERENCES:
- [Derived] Axelsson A, Iversen K, Vejlstrup N, Ho CY, Havndrup O, Kofoed KF, Norsk J, Jensen M, Bundgaard H. Functional effects of losartan in hypertrophic cardiomyopathy-a randomised clinical trial. Heart. 2016 Feb 15;102(4):285-91. doi: 10.1136/heartjnl-2015-308343. Epub 2015 Dec 9. PMID 26661322
- [Derived] Axelsson A, Iversen K, Vejlstrup N, Ho C, Norsk J, Langhoff L, Ahtarovski K, Corell P, Havndrup O, Jensen M, Bundgaard H. Efficacy and safety of the angiotensin II receptor blocker losartan for hypertrophic cardiomyopathy: the INHERIT randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2015 Feb;3(2):123-31. doi: 10.1016/S2213-8587(14)70241-4. Epub 2014 Dec 19. PMID 25533774